CLINICAL TRIAL: NCT00253331
Title: Phase III Laboratory Study of a Topical Gel Formulation of Nitroglycerin, MQX-503, in the Treatment of Raynaud's Phenomenon
Brief Title: Lab Study of MQX-503 in Treatment of Raynaud's
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: MQT 03-001
Record Dates: First submitted 2005-11-13; First posted 2005-11-15 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Raynaud Disease; Raynaud Disease Secondary to Scleroderma; Raynaud Secondary to Other Autoimmune Disease
Keywords: Raynaud's; sclerderma; systemic sclerosis; autoimmune disease
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic; Autoimmune Diseases | interventions — Nitroglycerin

INTERVENTIONS:
Drug: topical organogel with nitroglycerin

SUMMARY:
The purpose of this study is to determine, in comparison to a placebo control, the response to two dosage strengths of a topical gel formulation of nitroglycerin, MQX-303, in the determination of finger blood flow and skin temperature in the fingers of patients with moderate to severe Raynaud's phenomenon, follwoing exposure to cold temperatures.

Blood flow is determined by scanning laser Doppler equipment and skin temperature is measured using attached thermistor probes. Following baseline measurements, the study gel is applied, the hand is placed in a cold chamber, and then blood flow and skin temperature are monitored for the next two hours.

Each patient will receive multiple doses on different days so that each can serve as his/her own control in interpreting the response.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Raynaud's phenomenon
* outpoatients
* agree to apply gel as per protocol
* willing to discontinue current vasodilator therapy
* agree to stop other investigational medication for Raynaud's
* negative pregnancy test is fertile females
* able to give written informed consent and comply with study requirements

Exclusion Criteria:

* current use of ay nitrate medication or medications that interact with nitroglycerin
* patients with a known allergy to nitroglycerin or topical gel ingredients
* patients with a history of migraine headaches
* patients with unstable medical problems
* patients with cognitive or language difficulties
* patients with screening lab values more than 20% outside of normal
* patients with open lesions at site of application
* women of child-bearing potential who are unwilling to comply with contraceptive requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2004-11; Study Completion 2005-09

PRIMARY OUTCOMES:
Differntial time for blood flow to return to baseline following cold exposure.

SECONDARY OUTCOMES:
Differential time for skin temperature to return to baseline following cold exposure.
Quantitative reduction or prevention in symptoms following cold exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Hummers, MD, Principal Investigator — Johns Hopkins University; Carin Dugowson, MD, MPH, Principal Investigator — University of Washington Medical College
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - University of Washington Medical College, Seattle, Washington